CLINICAL TRIAL: NCT06124898
Title: Development and Initial Testing of a Multi-Component Breath Alcohol- Focused Intervention for Young Adults
Brief Title: Multi-Component Breath Alcohol Intervention
Acronym: BAMTECH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB22-11-43; R34AA029224-01 (NIH)
Record Dates: First submitted 2023-10-30; First posted 2023-11-09 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use; Alcohol Drinking; Drinking Behavior
MeSH Terms: conditions — Alcohol Drinking; Drinking Behavior | interventions — Motivational Interviewing; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate drinking technologies with "lower tech" facilitation (Experimental): Brief motivational-interviewing-based counseling followed by use of three moderate drinking technologies (breath alcohol device and app, blood alcohol content estimator app and self-texting procedure) with "lower tech" facilitation.
  Interventions: Device: Alcohol-related mobile health technologies; Behavioral: Motivational interview and psychoeducation on blood/breath alcohol concentration; Behavioral: Lower tech facilitation
- Moderate drinking technologies with "higher tech" facilitation (Experimental): Brief motivational-interviewing-based counseling followed by use of three moderate drinking technologies (breath alcohol device and app, blood alcohol content estimator app and self-texting procedure) with "higher tech" facilitation
  Interventions: Device: Alcohol-related mobile health technologies; Behavioral: Motivational interview and psychoeducation on blood/breath alcohol concentration; Device: Higher tech facilitation
- Attention control condition (Active Comparator): To be determined attention control condition, which will involve either non-personalized information about alcohol or feedback regarding another health behavior with minimal relationship to alcohol use, followed by related technology use.
  Interventions: Behavioral: Attention control psychoeducation; Device: Attention control technology

INTERVENTIONS:
Device: Alcohol-related mobile health technologies — Participants will be asked to use the three mobile technologies as they choose while drinking for a two-week period.
  Other Names: Smartphone breathalyzer, BAC estimator app and self-texting procedure
  Arms: Moderate drinking technologies with "higher tech" facilitation; Moderate drinking technologies with "lower tech" facilitation
Behavioral: Motivational interview and psychoeducation on blood/breath alcohol concentration — Brief 25/30-minute motivational interview and psychoeducation on blood/breath alcohol concentration that includes both personalized and standardized information.
  Other Names: M.I.
  Arms: Moderate drinking technologies with "higher tech" facilitation; Moderate drinking technologies with "lower tech" facilitation
Behavioral: Lower tech facilitation — Study staff will review instructions for technology use closely with participants and guide them in use of existing phone technologies as reminders for use of the three moderate drinking technologies during drinking situations.
  Arms: Moderate drinking technologies with "lower tech" facilitation
Device: Higher tech facilitation — Participants will use an app developed during the study that will provide protective behavioral strategies and reminders for use of the three moderate drinking technologies during drinking situations.
  Arms: Moderate drinking technologies with "higher tech" facilitation
Behavioral: Attention control psychoeducation — Brief 25/30-minute psychoeducation on a topic not related to alcohol use that will be developed in the course of the study.
  Arms: Attention control condition
Device: Attention control technology — App or other form of technology that will be developed in the course of the study to deliver information not related to alcohol use
  Arms: Attention control condition

SUMMARY:
This is the first stage of a three-stage, NIH-funded study to develop and test initially a multi-modal intervention concerning blood/breath alcohol concentration for young adults. The multimodal intervention will be made up of brief telehealth counseling and psychoeducation and use of three mobile technologies to facilitate moderate drinking. In the first stage of the study, we will conduct formative research to obtain input from the study population, test initially the telehealth version of the brief counseling and psychoeducation and to develop a simple, "low tech" approach to coaching participants to use the three mobile technologies in typical drinking situations. Participation will last approximately one month.

ELIGIBILITY:
Each subject must:

1. Be between the ages of 18-25
2. Be able to read English and complete study evaluations
3. Report at least four days with heavy episodic drinking (i.e., 4 or more drinks for women and 5 or more drinks for men) out of the prior 30 days
4. Report having consumed at least one alcoholic drink during a minimum of 12 days out of the prior 30 so that subjects will have multiple opportunities to use the moderate drinking technologies during the intervention period.
5. Meet, at minimum, DSM-5 criteria for a mild alcohol use disorder (i.e., meet at least 2 diagnostic criteria)
6. Self-report interest in using a smartphone app to help reduce drinking with a score of at least 3 on a 0-10 scale indicating at least a degree of openness to using technology to moderate drinking.

Exclusion Criteria

No subject may:

1. Have been in inpatient or intensive outpatient treatment within the past 12 months
2. Have used a smartphone application to facilitate moderate drinking more than 1 time within the past 12 months
3. Meet DSM-5 criteria for current substance use disorder with the exception of tobacco use disorder, mild or moderate alcohol use disorder or mild cannabis use disorder.
4. History of alcohol withdrawal or medically-assisted detoxification as individuals with this history will likely be in need of more intensive treatment than is offered in this study.
5. Be psychotic or otherwise severely psychiatrically disabled
6. Report a history of a medical condition that would contraindicate the consumption of alcohol (e.g., liver disease, cardiac abnormality, pancreatitis, diabetes, neurological problems, and gastrointestinal disorders)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Technology utilization | Across the field testing period, 2-4 weeks
  Percentage of reported drinking days on which one reports that moderate drinking technology use has occurred
Acceptability | At the end of the field testing period, 2-4 weeks
  Score on acceptability subscale of Modified System Usability Scale
Usability | At the end of the field testing period, 2-4 weeks
  Score on acceptability subscale of Modified System Usability Scale

SECONDARY OUTCOMES:
Drinks per drinking day | Across the field testing period, 2-4 weeks
  Number of drinks per day during field testing period
Estimated blood alcohol content | Across the field testing period, 2-4 weeks
  Average estimated blood alcohol content reached on drinking days
Negative consquences | At the end of the field testing period, 2-4 weeks
  Score on the Young Adult Alcohol Consequences Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Leeman, PhD., Principal Investigator — Northeastern University
Locations (1):
- EDGE Lab, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Study materials and datasets with identifiers removed will be shared with other investigators upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study materials are available at any time upon request. Datasets with identifiers removed will be available after publication of the main outcome paper from the study
Access Criteria: Any qualified investigator upon request